CLINICAL TRIAL: NCT01110252
Title: Unicentric Study Protocol of Cell Therapy in Chronic Obstructive Pulmonary Disease
Brief Title: Safety Study of Cell Therapy to Treat Chronic Obstructive Pulmonary Disease
Acronym: COPD-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Laboratório de Genética Humana e Terapia Celular, Unesp - Assis (Unknown); Instituto de Molestias Cardiovasculares (Other)
Responsible Party: Principal Investigator, João Tadeu Ribeiro Paes, sponsor, UPECLIN HC FM Botucatu Unesp
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: upeclin/ASSIS Unesp - 001
Record Dates: First submitted 2010-04-20; First posted 2010-04-26 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Emphysema
Keywords: Chronic Obstructive Pulmonary Disease; Emphysema; Cell therapy; Bone marrow mononuclear cells; stem cells
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pre-procedure (Active Comparator): emphysema patients evaluated prior to the stem cells infusion
  Interventions: Drug: Stem cells stimulation; Procedure: stem cells collection; Genetic: stem cells infusion
- post-procedure (Experimental): emphysema patients evaluated 30 days after the stem cells infusion
  Interventions: Drug: Stem cells stimulation; Procedure: stem cells collection; Genetic: stem cells infusion

INTERVENTIONS:
Drug: Stem cells stimulation — Subcutaneous injection of 5mcg/kg of G-CSF 3 days before the procedure.
  Other Names: Filgrastin - ACHÉ Laboratories.
Procedure: stem cells collection — pullout of 200ml of bone marrow through the puncture of the iliac crest
  Other Names: bone marrow harvest
Genetic: stem cells infusion — slow infusion through the brachial vein of 30ml of bone marrow mononuclear cells diluted in albuminous saline.
  Other Names: adult stem cell infusion

SUMMARY:
The purpose of this study is to determine whether the cell therapy with bone marrow mononuclear cells is safe in the treatment of chronic obstructive pulmonary disease, specifically the pulmonary emphysema.

DETAILED DESCRIPTION:
The main feature of the pulmonary emphysema, included in range of the Chronic Obstructive Pulmonary Disease (COPD), is the airflow obstruction resulting from the destruction of the alveolar walls distal to the terminal bronchiole, without significant pulmonary fibrosis. The existing clinical approaches has contributed to the enlargement and amelioration of the emphysema patients life quality, although no effective or curative treatment has been achieved. The surgical treatment, on the other hand, involves complex procedures and, in the specific case of lung transplantation, a lack of donors.

Considering these aspects, several experimental models have been proposed aiming to increase knowledge about the pathophysiological processes and enable new clinical approaches to the pulmonary emphysema. The cell therapy, briefly described as the use of cells in disease treatment, presents itself as a promising therapeutic approach with great potential applicability in degenerative pulmonary diseases. In this way, it is intended in this project, the proposition of a protocol to evaluate the safety of cell therapy with pool of mononuclear cells from bone marrow in patients with clinical and laboratory diagnosis of pulmonary emphysema in advanced stage (stage IV dyspnea).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe chronic obstructive pulmonary disease
* ineffective clinical treatment
* limited life expectancy
* limitations in daily physical activity
* possibility of pulmonary rehabilitation physiotherapy
* acceptable nutritional status
* acceptable cardiac function
* at least six months smoking cessation
* family support
* modified medical research council dyspnea scale stage > 3

Exclusion Criteria:

* pulmonary or extra-pulmonary infection
* severe coronary disease and/or ventricular dysfunction
* significant kidney or liver disease
* immunosuppressive disease
* active smoker
* cancer
* psychosocial problems
* established medical protocol
* family rejection
* pregnancy

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: João T Ribeiro-Paes, PhD MD, Principal Investigator — geneticist; Aldemir Bilaqui, MD, Study Director — surgeon; Oswaldo T Greco, MD, Study Chair — cardiologist; Milton A Ruiz, MD, Study Chair — hematologist; José D Araújo, MD, Study Chair — surgeon; Mario R Lago, Ms, Study Chair — technician
Locations (1):
- Laboratório de Genética Humana e Terapia Celular, Assis, São Paulo, Brazil

REFERENCES:
- [Derived] Ribeiro-Paes JT, Stessuk T, Marcelino M, Faria C, Marinelli T, Ribeiro-Paes MJ. A protocol proposition of cell therapy for the treatment of chronic obstructive pulmonary disease. Rev Port Pneumol. 2014 Mar-Apr;20(2):84-91. doi: 10.1016/j.rppneu.2013.06.008. Epub 2013 Nov 26. English, Portuguese. PMID 24287082
- [Derived] Ribeiro-Paes JT, Bilaqui A, Greco OT, Ruiz MA, Marcelino MY, Stessuk T, de Faria CA, Lago MR. Unicentric study of cell therapy in chronic obstructive pulmonary disease/pulmonary emphysema. Int J Chron Obstruct Pulmon Dis. 2011 Jan 1;6:63-71. doi: 10.2147/COPD.S15292. PMID 21311694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2009 to October 2009 four patients with clinical and laboratory diagnosis for advanced pulmonary emphysema were enrolled
Pre-assignment Details: Patients signed the Knowledge and Free Consent Instrument (TCLE)
Groups:
- Prior Then Post Procedure (Stem Cells Infusion): emphysema patients evaluated prior or after the infusion of the autologous stem cells
Period: Pre-procedure (Stem Cells Infusion)
Arm/Group | Prior Then Post Procedure (Stem Cells Infusion)
Started | 4
Completed | 4
Not Completed | 0
Period: Post-procedure (Stem Cells Infusion)
Arm/Group | Prior Then Post Procedure (Stem Cells Infusion)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prior Then Post Procedure (Stem Cells Infusion)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 65.75 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  Brazil | 4

OUTCOME MEASURES:

1. Primary Outcome: Forced Vital Capacity (FVC)
Description: A pulmonary function test that measures the volume and speed of the inhalated air.
Time Frame: baseline and 30 days after procedure
Population: all patients were evaluated prior and after the procedure
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Prior to the Procedure (Stem Cells Infusion): emphysema patients evaluated prior to the infusion of autologous stem cells
- Post Procedure (Stem Cells Infusion): emphysema patients evaluated 30 days after the infusion of autologous stem cells
Arm/Group | Prior to the Procedure (Stem Cells Infusion) | Post Procedure (Stem Cells Infusion)
Number analyzed (Participants) | 4 | 4
liters | 1.5 (0.2) | 2.1 (0.2)

2. Primary Outcome: Forced Expiratory Volume (FEV1)
Description: A pulmonary function test that measures the volume and speed of the exhaled air.
Time Frame: baseline and 30 days after procedure
Population: all patients were evaluated prior and after the procedure
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Prior to the Procedure (Stem Cells Infusion) | Post Procedure (Stem Cells Infusion)
Number analyzed (Participants) | 4 | 4
liters | 0.7 (0.1) | 0.8 (0.1)

3. Secondary Outcome: Arterial Blood Gases Test - Pa O2
Description: presence of oxygen in the blood gases.
Time Frame: baseline and 30 days after procedure
Population: all patients were evaluated prior and after the procedure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prior to the Procedure (Stem Cells Infusion) | Post Procedure (Stem Cells Infusion)
Number analyzed (Participants) | 4 | 4
mmHg | 69 (3) | 57 (3)

4. Secondary Outcome: Arterial Blood Gases Test - Pa CO2
Description: presence of CO2 in the arterial blood.
Time Frame: baseline and 30 days after the procedure
Population: all patients were evaluated prior and after the procedure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Prior to the Procedure (Stem Cells Infusion) | Post Procedure (Stem Cells Infusion)
Number analyzed (Participants) | 4 | 4
mm Hg | 48.75 (2.7) | 89.25 (2.7)

5. Primary Outcome: Vital Capacity - VC
Description: A pulmonary function test that measures the volume and speed of the inhalated and exhaled air.
Time Frame: baseline and 30 days after the procedure
Population: all patients were evaluated prior and after the procedure.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Prior to the Procedure (Stem Cells Infusion) | Post Procedure (Stem Cells Infusion)
Number analyzed (Participants) | 4 | 4
liters | 1.8 (0.3) | 1.4 (0.3)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Prior Then Post Procedure (Stem Cells Infusion)
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes